CLINICAL TRIAL: NCT07359092
Title: Comparison of Spexin and Phoenixin-20 Levels in Girls With Central Precocious Puberty, Premature Thelarche, and Healthy Controls
Brief Title: Spexin and Phoenixin-20 in Girls With Central Precocious Puberty
Acronym: SPX-PNX-CPP-20
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Serkan Bilge Koca, Associate Professor Dr, Kayseri City Hospital
Other Study IDs: SPX-PNX-CPP-2024
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Central Precocious Puberty (CPP); Puberty Disorders; Puberty; Hypothalamic-Pituitary-Ovarian Axis Dysfunction (Disorder)
Keywords: Spexin; Phoenixin-20; Children; Girls; Puberty; Precocious puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Central Precocious Puberty (CPP): Girls younger than 8 years diagnosed with CPP based on clinical findings (breast development stage) and LH-RH stimulation test peak LH level >5 mIU/mL
- Premature Thelarche (PT): Girls younger than 8 years presenting with isolated breast development and LH-RH stimulation test peak LH level <5 mIU/mL
- Healthy controls: Age-matched healthy girls without signs of breast development

SUMMARY:
Central precocious puberty (CPP) is characterized by the early activation of the hypothalamic-pituitary-gonadal axis in girls and may be difficult to distinguish from benign variants such as premature thelarche. Spexin and phoenixin-20 are novel neuropeptides that have been suggested to play roles in reproductive axis regulation.

The aim of this study was to compare serum spexin and phoenixin-20 levels among girls with central precocious puberty, girls with premature thelarche, and healthy age-matched controls. The study evaluated whether these biomarkers could help differentiate CPP from other conditions presenting with early breast development.

Clinical, anthropometric, and biochemical parameters were analyzed in all participants. Blood samples were collected and serum spexin and phoenixin-20 levels were measured using commercially available assay kits.

DETAILED DESCRIPTION:
This was a prospective, observational study conducted in a pediatric endocrinology outpatient clinic. The study population consisted of girls younger than 8 years of age who presented between December 2024 and December 2025. Participants were categorized into three groups: girls diagnosed with central precocious puberty (CPP), girls with premature thelarche (PT), and healthy age-matched control subjects. The CPP group: 33 patients, PT group: 57 patients, and healthy controls: 53 patients.

The diagnosis of central precocious puberty was based on clinical findings, auxological data, bone age assessment, and hormonal evaluation according to standard pediatric endocrinology criteria. Premature thelarche was defined as isolated breast development without other signs of pubertal progression or activation of the hypothalamic-pituitary-gonadal axis.

Clinical and anthropometric data, including age, height, weight, body mass index, bone age, were recorded. Blood samples were obtained under standardized conditions, and also LH-RH stimulation test was applied in CPP and PT groups. Basal and stimulated FSH and LH hormone levels were examined. In addition, serum spexin and phoenixin-20 concentrations were measured using enzyme-linked immunosorbent assay kits in accordance with the manufacturers' instructions.

The primary objective of the study was to investigate whether serum spexin and phoenixin-20 levels differ between girls with CPP and those with PT or healthy controls, and whether these biomarkers could aid in distinguishing CPP from other causes of early pubertal signs.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age younger than 8 years,
* Presentation for evaluation of early pubertal signs (breast development)
* Classification into one of the following groups: central precocious puberty, premature thelarche, or healthy control

Exclusion Criteria:

* Presence of peripheral precocious puberty,
* Known chronic systemic disease,
* Use of medications affecting the hypothalamic-pituitary-gonadal axis,
* Known genetic syndromes of congenital endocrine disorders

Ages: 4 Years to 8 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female only
Study Population: Girls younger than 8 years who presented for evaluation of early pubertal signs between December 2024 and December 2025. Participants were classified into two groups: CPP and PT; according to LH-RH stimulation test peak LH levels. And a third group was included (totally three groups) for age matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Serum Spexin and Phoenixin-20 levels | At initial clinical evaluation
  Comparison of serum Spexin and Phoenixin-20 concentrations among girls with central precocious puberty, premature thelarche, and healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared from this study